CLINICAL TRIAL: NCT02473133
Title: Randomized Phase II-III Study of Personalized Radiotherapy Dose Redistribution in Patients With Inoperable Stage III Non-small Cell Lung Cancer and a Persistent FDG Uptake at 42 Grays During Concomitant Radio-chemotherapy
Brief Title: Study of Interest of Personalized Radiotherapy Dose Redistribution in Patients With Stage III NSCLC
Acronym: RTEP7
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Collaborators: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHB14.04/IFCT14-02
Record Dates: First submitted 2015-06-08; First posted 2015-06-16 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: radiotherapy; dose redistribution; boost
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Personalized dose redistribution (Experimental): Patients in the will receive an individualized radiotherapy prescription up to a total dose of 74 Gy given in 6.6 weeks if they have a positive FDG-PET at 42Gy (about two thirds of patients are expected as positive). An initial dose of 50 Gy will be delivered in 5 weeks (single daily fractions of 2 Gy), then an additional dose up to 24 Gy will be delivered over 1.6 week using a twice-a-day fractionated radiotherapy.
  Interventions: Radiation: Personalized dose redistribution
- No dose redistribution (Sham Comparator): Patients will receive a single prescription of 66 Gy in 33 fractions in 6.6 weeks, with 2 Gy fractions given once daily, 5 days a week, without target volume reduction or adaptation (whatever the FDG-PET result).
  Interventions: Radiation: No personalized dose redistribution

INTERVENTIONS:
Radiation: Personalized dose redistribution — Patients will receive an individualized radiotherapy prescription up to a total dose of 74 Gy given in 6.6 weeks if they have a positive FDG-PET at 42Gy. An initial dose of 50 Gy will be delivered in 5 weeks (single daily fractions of 2 Gy), then an additional dose up to 24 Gy will be delivered over 1.6 week.
  Other Names: boost
  Arms: Personalized dose redistribution
Radiation: No personalized dose redistribution — Patients will receive a single prescription of 66 Gy in 33 fractions in 6.6 weeks, with 2 Gy fractions given once daily, 5 days a week, without target volume reduction or adaptation (whatever the FDG-PET2 result).
  Arms: No dose redistribution

SUMMARY:
In patients with locally advanced stage III non-small cell lung cancer, the probability of local control remains low (about 17% at 1 year). Concomitant radio-chemotherapy is the standard treatment. An increase in total radiotherapy dose (from 66 to 74 Gray) has been proposed to improve local control, with contradictory results.

Relevant FDG-PET scan images can be acquired during radio-chemotherapy, with a demonstrated prognostic impact and recently in a multicentre prospective study. A significant reduction in FDG uptake / volume (metabolic response) suggests that the radiotherapy target volume could be reduced during radiotherapy possibly improving organs at risk tolerance. Conversely, a lack of metabolic response may justify treatment intensification before the end of radiotherapy. The investigators hypothesis is to investigate the individual tumour heterogeneity on FDG-PET during radio-chemotherapy to reduce the volume to a biological target that could receive a higher total dose (personalized dose redistribution).

DETAILED DESCRIPTION:
The investigators objective is to determine whether tumour radiotherapy dose escalated up to 74 Gy in 6.6 weeks can improve the disease Local Regional Control rate at 15 months (1 year after completion of RCT) by adapting radiotherapy target volume to the metabolic response as assessed on FDG-PET/CT performed at 42 Gy of concomitant radio-chemotherapy in stage III non-small cells lung cancer and warrant more extensive phase III study.

Eligible patients will be allocated to one of 2 treatment groups:

* Arm A: Patients in the experimental arm will receive an individualized radiotherapy prescription up to a total dose of 74 Gy given in 6.6 weeks if they have a positive FDG-PET at 42Gy.
* Arm B: Patients in the standard arm will receive a single prescription of 66 Gy in 33 fractions in 6.6 weeks, with 2 Gy fractions given once daily, 5 days a week, without target volume reduction or adaptation (whatever the FDG-PET result).

In both arms, all patients will undergo 2 cycles of induction chemotherapy (based platinum salts) and a curative radio-chemotherapy. In both arms all fields must be treated daily.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients,
* Age over 18 years and below 75-year-old,
* Good general condition: WHO performance status ≤ 1,
* Histological evidence of non-small cell lung cancer,
* Measureable tumour according to RECIST 1.1 evaluation criteria,
* Mediastinoscopy or endobronchial ultrasound to prove the histological stage N2/N3,
* Patient eligible to curative-intent radio-chemotherapy,
* Absence of pleural involvement, of pulmonary or extra-thoracic metastatic localisation,
* Absence of co-morbidity contra-indicating radio-chemotherapy,
* Lung function: FEV1 ≥ 40% of theoretical value and DLCO/VA ≥ 60% of theoretical value and PaO2 ≥ 60 mm Hg,
* Tumour FDG uptake higher than mediastinal background noise on baseline PET/CT,
* Haematological parameters:
* Neutrophil count ≥ 1.5x109/L and platelet count ≥ 100x109/L,
* Haemoglobin ≥ 9 g/dL,
* Provisional RT plan confirming that the dose objectives (minimal dose of 62.7 Gy (95% of the prescribed dose) in 98% of target volumes and 70.3 Gy for the "boosted" volume at 74 Gy) and constraints (lungs, spinal cord) are met (ICRU83),
* Estimated creatinine clearance ≥ 60 mL/min,
* Signed informed consent
* Affiliated or beneficiary of a social benefit system

Exclusion Criteria:

* Histology other than non-small cell lung cancer,
* Absence of FDG uptake on FDG-PET/CT scan before induction chemotherapy,
* Patients for whom curative radiotherapy is not indicated (tumour extension, metastases, general condition, co-morbidities),
* Significant interstitial disease on CT scan,
* Previous neoplastic disease of less than 5 years duration or progressive (without basal cell carcinoma of the skin, in situ carcinoma of the cervix),
* Previous thoracic radiotherapy,
* Patient enrolled in another therapeutic trial,
* Pregnant women or women of child-bearing potential or breast feeding mothers,
* Adult subjects who are under protective custody or guardianship,
* Patient unable to comply with the specific obligations of the study (geographic, social or physical reasons),
* Uncontrolled diabetes with blood glucose ≥10 mmol/L,
* Hypersensitivity to the active substance (FDG) or to any of the excipients,
* Patients unable to understand the purpose of the study (language, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2015-11-12 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Local regional control rate | one year
  LCR rate (responders or stable disease) at 1 year after completion of RCT (M15 visit). Disease progression will be assessed by RECIST 1.1 criteria

SECONDARY OUTCOMES:
Percentage of local regional control with RECIST 1.1 criteria | assessed at 9 months, 15 months, 27 months and 39 months
  Disease progression will be assessed by RECIST 1.1 criteria
interval from the date of registration to date of local or regional progression | 3 years
  the interval from the date of registration to date of local or regional progression
Percentage of severe (grade 3+ CTCAE, v4) radiation-induced toxicity affecting lung and oesophagus at M9 visit (early toxicity) and M15, M27, M39 visits (late toxicity), | assessed at 9 months, 15 months, 27 months and 39 months
  Percentage of severe (grade 3+ CTCAE, v4) radiation-induced toxicity affecting lung and oesophagus at M9 visit (early toxicity) and M15, M27, M39 visits (late toxicity),
Percentage of patients in arm A for whom the radiotherapy dose could be increased | 6.6 weeks
  Percentage of patients in arm A for whom the RT dose could be increased
correlation of progression free survival with PET measure | one year
  standardized uptake value max and metabolic tumor volume of FDG -PET2 will be correlated with progression free survival at M15 visit
correlation of overall survival with PET measure | one year
  standardized uptake value max and metabolic tumor volume of FDG -PET2 will be correlated with overall survival at M15 visit
Change in standardized uptake value max | weeks 12
  Measurements of the relative change in SUVmax from the 18F-FDG -PET1 (baseline) to the FDG -PET2 at 42 Gy defined as [(PET2- PET1) / PET1] x 100%
Change in metabolic volume | weeks 12
  Measurements of the relative change metabolic tumour volume from the 18F-FDG -PET1 (baseline) to the FDG -PET2 at 42 Gy defined as [(PET2- PET1) / PET1] x 100%
Overall Survival | assessed at 9 months, 15 months, 27 months and 39 months
  overall survival after M9, M15, M27, M39 follow-up visits
progression-free survival | assessed at 9 months, 15 months, 27 months and 39 months
  progression-free survival after M9, M15, M27, M39 follow-up visits

CONTACTS AND LOCATIONS:
Overall Officials: Peirre Vera, MD,PHD, Principal Investigator — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France

REFERENCES:
- [Derived] Vera P, Thureau S, Le Tinier F, Chaumet-Riffaud P, Hapdey S, Kolesnikov-Gauthier H, Martin E, Berriolo-Riedinger A, Pourel N, Broglia JM, Boissellier P, Guillemard S, Salem N, Brenot-Rossi I, Le Pechoux C, Berthold C, Giroux-Leprieur E, Moreau D, Guillerm S, Benali K, Tessonnier L, Audigier-Valette C, Lerouge D, Quak E, Massabeau C, Courbon F, Moisson P, Larrouy A, Modzelewski R, Gouel P, Ghazzar N, Langlais A, Amour E, Zalcman G, Giraud P. Adaptive radiotherapy (up to 74 Gy) or standard radiotherapy (66 Gy) for patients with stage III non-small-cell lung cancer, according to [18F]FDG-PET tumour residual uptake at 42 Gy (RTEP7-IFCT-1402): a multicentre, randomised, controlled phase 2 trial. Lancet Oncol. 2024 Sep;25(9):1176-1187. doi: 10.1016/S1470-2045(24)00320-6. Epub 2024 Aug 9. PMID 39134086